CLINICAL TRIAL: NCT04528069
Title: Clinical Investigation of the Visual Outcomes and Safety of AcrySof® IQ PanOptix® Toric Trifocal IOLs in an Asian Population
Brief Title: Clinical Investigation of the Visual Outcomes and Safety of a Trifocal Toric IOL in an Asian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX140-P001
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-01

CONDITIONS: Aphakia; Corneal Astigmatism
Keywords: Intraocular lens; Cataract
MeSH Terms: conditions — Aphakia; Astigmatism; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PanOptix Toric Trifocal IOL (Experimental): PanOptix Toric Trifocal IOL implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient. Both eyes will be implanted (bilateral implantation).
  Interventions: Device: ACRYSOF® IQ PanOptix® Toric Trifocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: ACRYSOF® IQ PanOptix® Toric Trifocal IOL — Single-piece, ultraviolet and blue-light filtering, foldable, multifocal toric IOL intended to provide vision to aphakic subjects at near, intermediate, and distance and to correct pre-existing corneal astigmatism. This device is approved in Australia.
  Other Names: PanOptix Toric Trifocal IOL; Models TFNT30, TFNT40, TFNT50, TFNT60
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation of the IOL per investigator's standard of care and instructions for use

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the ACRYSOF® IQ PanOptix® Toric Trifocal intraocular lens (IOL) when implanted in the eye following cataract removal in an Asian population.

DETAILED DESCRIPTION:
Both eyes will be implanted with the PanOptix Toric Trifocal IOL. The eye with the highest astigmatism will be implanted first. The second eye will be implanted within 7-14 days of the first eye.

Subjects will attend a total of 10 scheduled visits as follows: 1 screening visit, 1 operative visit for each eye, 2 post-operative visits for each eye, and 3 postoperative visits where both eyes will be evaluated. The duration of participation for each subject will be approximately 8 months.

This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Planned bilateral cataract removal followed by posterior chamber IOL implantation with PanOptix Toric (TFNT30, TFNT40, TFNT50, or TFNT60);
* Calculated target residual refractive error within ±0.50 diopter (D) of emmetropia within the commercially available IOL Power Range in both operative eyes;
* Preoperative regular corneal keratometric astigmatism with predicted residual refractive astigmatism ≤ 0.50 diopter (D) in both operative eyes;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Preoperative irregular astigmatism;
* Clinically significant corneal abnormalities;
* Glaucoma;
* History of or current retinal disease; anterior or posterior segment inflammation;
* Other planned ocular surgical procedures including, but not limited to, limbal relaxing incision (LRI)/Astigmatic Keratotomy and laser-assisted in situ keratomileusis (LASIK);
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (4):
- Australia (4):
  - Alcon Investigator 8117, Campsie, New South Wales
  - Alcon Investigator 7678, Sydney, New South Wales
  - Alcon Investigator 7813, Footscray, Victoria
  - Alcon Investigator 8122, Saint Albans, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigative sites located in Australia.
Pre-assignment Details: A total of 58 subjects were enrolled in the study (i.e., signed informed consent), of whom 4 were screen failures. This reporting group includes all subjects (54) implanted with the IOL in one or both eyes.
Units Other Than Participants: eyes
Groups:
- PanOptix Toric Trifocal IOL: PanOptix Toric Trifocal intraocular lens (IOL) implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient. Both eyes were implanted (bilateral implantation).
Period: Overall Study
Arm/Group | PanOptix Toric Trifocal IOL
Started | 54; 105 eyes
First Eye Implanted | 54; 54 eyes
Second Eye Implanted | 51; 51 eyes
Completed | 50; 97 eyes
Not Completed | 4; 8 eyes
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Patient Unable to Come | 1
Not completed — Patient Unable to Attend | 1

BASELINE CHARACTERISTICS:
Population: All Implanted Analysis Set: All eyes with successful IOL implantation with at least one post-operative visit
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0
  Black or African American | 0
  American Indian or Alaska Native | 0
  Asian | 54
  Native Hawaiian or Other Pacific Islander | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  Australia | 54
Specific Asian Nationality [Count of Participants; unit: Participants]
  Chinese | 54
  Japanese | 0
  Korean | 0
  Mongolian | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Monocular Residual Manifest Cylinder for All Operative Eyes for All IOL Models Combined
Description: Manifest cylinder is the amount of added correction needed to compensate for any astigmatism that may be present. A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Residual manifest cylinder was measured in diopters and reported in plus cylinder form, with a smaller number indicating a lesser amount of added correction. Eyes were assessed individually and combined for the analysis. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Month 3 postoperative, Month 6 postoperative
Population: All-Implanted Analysis Set (AAS): All eyes with successful IOL implantation with at least one post-operative visit and data at study visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Groups:
- All Eyes: PanOptix Toric Trifocal intraocular lens (IOL) implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient
Arm/Group | All Eyes
Number analyzed (Participants) | 50
Number analyzed (eyes) | 98
diopter
  Month 3 postoperative | 0.219 (0.2388)
  Month 6 postoperative: number analyzed (eyes) | 97
  Month 6 postoperative | 0.198 (0.2392)

2. Primary Outcome: Percentage of Eyes With IOL Rotation Less Than 10 Degrees
Description: IOL rotation was defined as the difference in IOL axis of orientation from Day 1 postoperative. IOL rotation was assessed by the investigator using a slit lamp and was recorded in degrees, with a smaller number indicating less rotation. Eyes were assessed individually and combined for the analysis. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Month 3 postoperative, Month 6 postoperative
Population: AAS
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | All Eyes
Number analyzed (Participants) | 50
Number analyzed (eyes) | 98
percentage of eyes
  Month 3 postoperative | 100
  Month 6 postoperative: number analyzed (eyes) | 97
  Month 6 postoperative | 100

3. Primary Outcome: Mean Binocular Best Corrected Distance Visual Acuity (BCDVA)
Description: Visual acuity (VA) was assessed at a distance of 4 meters with refractive correction in place using a visual acuity chart. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.0 logMAR corresponding to 20/20 Snellen visual acuity, or normal distance eyesight. Eyes were assessed binocularly (eyes together). A lower value denotes better visual acuity. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Month 3 postoperative, Month 6 postoperative
Population: AAS
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- PanOptix Toric Trifocal IOL: PanOptix Toric Trifocal IOL implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient. Both eyes were implanted (bilateral implantation).
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 48
logMAR
  Month 3 postoperative | 0.043 (0.0881)
  Month 6 postoperative: number analyzed (Participants) | 47
  Month 6 postoperative | 0.022 (0.0810)

4. Primary Outcome: Mean Binocular Distance Corrected Intermediate Visual Acuity (DCIVA)
Description: Visual acuity (VA) was assessed at a distance of 60 meters with distance correction (plus or minus power) in place. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.0 logMAR corresponding to 20/20 Snellen visual acuity, or normal distance eyesight. Eyes were assessed binocularly (eyes together). A lower value denotes better visual acuity. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Month 3 postoperative, Month 6 postoperative
Population: AAS
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 48
logMAR
  Month 3 postoperative | 0.075 (0.1068)
  Month 6 postoperative: number analyzed (Participants) | 47
  Month 6 postoperative | 0.089 (0.1074)

5. Primary Outcome: Mean Binocular Distance Corrected Near Visual Acuity (DCNVA)
Description: Visual acuity (VA) was assessed at a distance of 40 centimeters with distance correction (plus or minus power) in place using a visual acuity chart. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.0 logMAR corresponding to 20/20 Snellen visual acuity, or normal distance eyesight. Eyes were assessed binocularly (eyes together). A lower value denotes better visual acuity. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Month 3 postoperative, Month 6 postoperative
Population: AAS
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 48
logMAR
  Month 3 postoperative | 0.161 (0.0924)
  Month 6 postoperative: number analyzed (Participants) | 47
  Month 6 postoperative | 0.139 (0.0886)

6. Primary Outcome: Percentage of Eyes With Secondary Surgical Interventions (SSIs), by Category
Description: A secondary surgical intervention (SSI) was defined as a surgical procedure occurring after primary implantation of the IOL. SSIs are reported categorically as SSIs related to the IOL and due to optical properties, SSIs related to the IOL and not due to optical properties, and SSIs unrelated to the IOL.
Time Frame: Up to Month 6 postoperative
Population: Safety Analysis Set (SAS): All eyes with attempted IOL implantation, successful or aborted after contact with the eye, and data at study visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- PanOptix Toric Trifocal IOL - First Eye; PanOptix Toric Trifocal IOL - Second Eye; PanOptix Toric Trifocal IOL - All Eyes: PanOptix Toric Trifocal intraocular lens (IOL) implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient
Arm/Group | PanOptix Toric Trifocal IOL - First Eye | PanOptix Toric Trifocal IOL - Second Eye | PanOptix Toric Trifocal IOL - All Eyes
Number analyzed (Participants) | 54 | 51 | 105
Number analyzed (eyes) | 54 | 51 | 105
percentage of eyes
  SSIs Related to IOL - Due to Optical Properties | 0.0 | 0.0 | 0.0
  SSIs Related to the IOL - Not Due to Optical Properties | 0.0 | 0.0 | 0.0
  SSIs Unrelated to the IOL | 1.9 | 2.0 | 1.9

7. Primary Outcome: Percentage of Subjects With a Severe Visual Disturbance
Description: The Questionnaire for Visual Disturbances (QUVID) is a patient-reported outcomes questionnaire that collects responses from the subject about 7 vision-related experiences. For each experience, the subject was asked if he/she had experienced it during the past 7 days. Subjects responding "Yes" were then asked to rate how severe their worst experience was during the past 7 days. Subjects responded on a 5-point scale: 0=None; 1=A little; 2=Mild; 3=Moderate; 4=Severe. Subjects responding "No" were automatically imputed as reporting, "0=None." Percentage was calculated as number of subjects with response in specified category divided by number of subjects with data regardless of response, times 100. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Preoperative, Month 3 postoperative, Month 6 postoperative
Population: SAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PanOptix Toric Trifocal IOL - Preoperative: Prior to attempted implantation with the PanOptix Toric Trifocal IOL
- PanOptix Toric Trifocal IOL - Month 3; PanOptix Toric Trifocal IOL - Month 6: PanOptix Toric Trifocal IOL implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient. Both eyes were implanted (bilateral implantation).
Arm/Group | PanOptix Toric Trifocal IOL - Preoperative | PanOptix Toric Trifocal IOL - Month 3 | PanOptix Toric Trifocal IOL - Month 6
Number analyzed (Participants) | 51 | 48 | 47
percentage of participants
  Starbursts - Severe: number analyzed (Participants) | 51 | 47 | 47
  Starbursts - Severe | 11.8 [4.4 to 23.9] | 17.0 [7.6 to 30.8] | 14.9 [6.2 to 28.3]
  Halos - Severe | 9.8 [3.3 to 21.4] | 6.3 [1.3 to 17.2] | 0.0 [0.0 to 7.5]
  Glare - Severe: number analyzed (Participants) | 51 | 48 | 46
  Glare - Severe | 19.6 [9.8 to 33.1] | 8.3 [2.3 to 20.0] | 6.5 [1.4 to 17.9]
  Hazy Vision - Severe | 9.8 [3.3 to 21.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]
  Blurred Vision - Severe: number analyzed (Participants) | 50 | 48 | 47
  Blurred Vision - Severe | 18.0 [8.6 to 31.2] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]
  Double Vision - Severe | 2.0 [0.0 to 10.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]
  Dark Area - Severe | 2.0 [0.0 to 10.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]

8. Primary Outcome: Percentage of Subjects With a Most Bothersome Visual Disturbance (QUVID)
Description: QUVID is a patient-reported outcomes questionnaire that collects responses from the subject about 7 vision-related experiences. For each experience, the subject was asked if he/she had experienced it during the past 7 days. Subjects responding "Yes" were then asked to rate how severe their worst experience was with the vision-related experience in the past 7 days. Subjects responded on a 5-point scale: 0=Not bothered at all; 1=Bothered a little bit; 2=Bothered somewhat; 3=Bothered quite a bit; 4=Bothered very much. Subjects responding "No" were automatically imputed as reporting, "0=Not bothered at all. Percentage was calculated as number of subjects with response in specified category divided by number of subjects with data regardless of response, times 100. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Preoperative, Month 3 postoperative, Month 6 postoperative
Population: SAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PanOptix Toric Trifocal IOL - Preoperative; PanOptix Toric Trifocal IOL - Month 3; PanOptix Toric Trifocal IOL - Month 6: PanOptix Toric Trifocal IOL implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient. Both eyes were implanted (bilateral implantation).
Arm/Group | PanOptix Toric Trifocal IOL - Preoperative | PanOptix Toric Trifocal IOL - Month 3 | PanOptix Toric Trifocal IOL - Month 6
Number analyzed (Participants) | 51 | 48 | 47
percentage of participants
  Starbursts - Bothered very much | 9.8 [3.3 to 21.4] | 4.2 [0.5 to 14.3] | 2.1 [0.1 to 11.3]
  Halos - Bothered very much | 7.8 [2.2 to 18.9] | 0.0 [0.0 to 7.4] | 2.1 [0.1 to 11.3]
  Glare - Bothered very much | 21.6 [11.3 to 35.3] | 6.3 [1.3 to 17.2] | 0.0 [0.0 to 7.5]
  Hazy Vision - Bothered very much | 13.7 [5.7 to 26.3] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]
  Blurred Vision - Bothered very much: number analyzed (Participants) | 50 | 48 | 47
  Blurred Vision - Bothered very much | 20.0 [10.0 to 33.7] | 2.1 [0.1 to 11.1] | 2.1 [0.1 to 11.3]
  Double Vision - Bothered very much | 5.9 [1.2 to 16.2] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]
  Dark Area - Bothered very much | 3.9 [0.5 to 13.5] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.5]

9. Primary Outcome: Percentage of Subjects With Ocular Serious Adverse Events Including Serious Adverse Device Effects
Description: An adverse event (AE) was defined as untoward medical occurrence, unintended disease or injury, or untoward clinical sign (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. No formal statistical hypothesis testing was prespecified for this outcome measure.
Time Frame: Up to Month 6 postoperative
Population: SAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PanOptix Toric Trifocal IOL - First Eye | PanOptix Toric Trifocal IOL - Second Eye
Number analyzed (Participants) | 54 | 51
percentage of participants
  Diabetic retinal oedema | 1.9 [0.5 to 9.89] | 0.0 [0.0 to 6.98]
  Intra-ocular injection | 1.9 [0.5 to 9.89] | 0.0 [0.0 to 6.98]
  Iris adhesions | 0.0 [0.0 to 6.60] | 2.0 [0.05 to 10.45]

10. Primary Outcome: Percentage of Subjects With Nonocular Serious Adverse Events Including Serious Adverse Device Effects
Description: as for outcome 9
Time Frame: Up to Month 6 postoperative
Population: SAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PanOptix Toric Trifocal IOL: PanOptix Toric Trifocal intraocular lens (IOL) implanted in the capsular bag in the posterior chamber following cataract surgery and intended for long-term use over the lifetime of the cataract patient
Arm/Group | PanOptix Toric Trifocal IOL
Number analyzed (Participants) | 54
percentage of participants
  Coronary arterial stent insertion | 1.9 [0.05 to 9.89]
  Coronary artery disease | 1.9 [0.05 to 9.89]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to Day 180-210 post-treatment/study exit, up to 8 months. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: This analysis population includes all eyes with attempted IOL implantation (successful or aborted after contact with the eye). "At Risk" population of pre-treatment and systemic AEs is reported in units of subjects; ocular AE population is reported in units of eyes.
Groups:
- Pretreatment: Events reported in this group occurred prior to attempted implantation with the test article
- PanOptix Toric First Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the first implanted eye
- PanOptix Toric Second Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the second implanted eye
- PanOptix Toric Systemic: Events reported in this group occurred after attempted implantation with the test article
Arm/Group | Pretreatment | PanOptix Toric First Eye | PanOptix Toric Second Eye | PanOptix Toric Systemic
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/54 | 1/51 | 1/54
Other Adverse Events (participants affected / at risk) | 0/54 | 5/54 | 4/51 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=54) | PanOptix Toric First Eye (N=54) | PanOptix Toric Second Eye (N=51) | PanOptix Toric Systemic (N=54)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iris adhesions (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-ocular injection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=54) | PanOptix Toric First Eye (N=54) | PanOptix Toric Second Eye (N=51) | PanOptix Toric Systemic (N=54)
Corneal erosion (Eye disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04528069/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT04528069/SAP_001.pdf